CLINICAL TRIAL: NCT03245853
Title: Epithelium-On Corneal Collagen Crosslinking for Keratoconus
Brief Title: Epi-On Corneal Crosslinking for Keratoconus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Comprehensive EyeCare of Central Ohio (Other)
Collaborators: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170265
Record Dates: First submitted 2017-08-09; First posted 2017-08-10 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Keratoconus; Keratoconus, Unstable
Keywords: Keratoconus; Corneal Crosslinking; CXL
MeSH Terms: conditions — Keratoconus | interventions — Flavin Mononucleotide

STUDY DESIGN:
Intervention Model Description: Subjects with a diagnosis of progressive keratoconus will be evaluated for suitability as a candidate for CXL. Subjects that are candidates for CXL will be asked to participate in this study and will undergo required screening testing. Informed consent will be obtained from each subject prior to study-oriented testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Other): Treatment as per protocol, there is no placebo arm.
  Interventions: Drug: Riboflavin 5'-Phosphate

INTERVENTIONS:
Drug: Riboflavin 5'-Phosphate — Photrexa (riboflavin 5'-phosphate ophthalmic solution) 0.146%, is a yellow sterile buffered solution containing 1.46 mg/mL riboflavin 5'-phosphate, The pH of the solution is approximately 7.1 and the osmolarity is 157-177 mOsm/kg. Each 1 mL of the solution contains 1.53 mg of riboflavin 5'-phosphate sodium (equivilant to 1.20 mg [0.12%] riboflavin). Riboflavin 5'-phosphate sodium USP is a mixture of the sodium salts of riboflavin, riboflavin monophosphates, and riboflavin diphosphates. The inactive ingredients are dibasic sodium phosphate, monbasic sodium phosphate, sodium chloride, and water for injection.
  Other Names: Photrexa

SUMMARY:
Epithelium-On Corneal Crosslinking for Keratoconus.

DETAILED DESCRIPTION:
Subjects with a diagnosis of progressive keratoconus will be evaluated for suitability as a candidate for Corneal Crosslinking (CXL). Subjects that as candidates for CXL will be asked to participate in this study and will undergo the required screening procedures to determine study eligibility. Informed consent will be obtained from each subject before performance of any required any required study procedures that are not part of the investigator's routine examination. All Subjects will be evaluated at screening/baseline, Day 0 (treatment day), then 1 day, 1 week, and 1, 3, 6, 12 months after treatment. Pentacam measurements and measurements of best spectacle-corrected visual acuity will be obtained and baseline and at appropriate times after the epithelium-on CXL procedure. Safety monitoring throughout the study will include observations at appropriate times for adverse events, clinically significant findings on ophthalmic examination, and slit-lamp examination.

The primary efficacy parameter is the change from baseline over time in maximum keratometry (K-Max). Addition analyses for efficacy will include uncorrected visual acuity (UCVA) and best corrected visual acuity (BCVA).

ELIGIBILITY:
Inclusion Criteria:

* 12 to 40 years of age, having a diagnosis of keratoconus, signed written informed consent, willingness and ability to comply with schedule for follow-up visits

Exclusion Criteria:

* Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications (herpes simplex/zoster, recurrent corneal erosion syndrome, corneal melt, corneal dystrophy, etc.) Pregnancy, intent to become pregnant, or lactation during study. Corneal pachymetry <350 microns at the thinnest point measured by Pentacam in the eye(s) to be treated.

Nystagmus or any other condition that would prevent steady gaze. Other systemic condition that in the investigator's opinion would not allow the patient to be a good candidate for the study.

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum keratometric change | 12 months
  Change from baseline keratometric maximum over time.

SECONDARY OUTCOMES:
Visual acuity change | 12 months
  Change from baseline uncorrected distance visual acuity and best spectacle-corrected visual acuity.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Beckman, M.D., Principal Investigator — Comprehensive EyeCare of Central Ohio
Locations (1):
- Comprehensive EyeCare of Central Ohio, Westerville, Ohio, United States

DOCUMENTS (2):
  • Study Protocol (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT03245853/Prot_000.pdf
  • Informed Consent Form (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT03245853/ICF_001.pdf